CLINICAL TRIAL: NCT00082316
Title: A Randomized, Open-Label Study of the Tolerability of Three Local Anesthetic Formulations in Conjunction With NGX-4010 for the Treatment of Neuropathic Pain
Brief Title: Tolerability of Three Local Anesthetic Formulations in Conjunction With NGX-4010 for the Treatment of Neuropathic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NeurogesX (Industry)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: C111
Record Dates: First submitted 2004-05-05; First posted 2004-05-07 (Estimated); Last update posted 2008-01-11 (Estimated); Status verified 2008-01

CONDITIONS: Herpes Zoster; Neuralgia; Pain; HIV Infections; Peripheral Nervous System Diseases; Diabetic Neuropathies; Diabetes Mellitus; Polyneuropathies
Keywords: Dermal assessment; Pain assessment; Diary; Analgesics; Capsaicin; Herpes zoster; Neuralgia; HIV Infections; Peripheral Nervous System Diseases; Diabetic Neuropathies; Diabetes Mellitus; Polyneuropathies; Complementary Therapies
MeSH Terms: conditions — Herpes Zoster; Neuralgia; Pain; HIV Infections; Peripheral Nervous System Diseases; Diabetic Neuropathies; Diabetes Mellitus; Polyneuropathies

INTERVENTIONS:
Drug: Capsaicin Dermal Patch

SUMMARY:
This study is a randomized, open-label multi-center evaluation of the tolerability of treatment with NGX-4010 in conjunction with pre-patch topical application of one of three 4% lidocaine-based local anesthetic products. Eligible subjects will have moderate to severe neuropathic pain secondary to painful diabetic neuropathy (PDN), postherpetic neuralgia (PHN) or HIV-associated neuropathy (HIV-AN), with average numeric pain rating scale (NPRS) scores during screening of 3 to 8 (inclusive).

ELIGIBILITY:
Key Eligibility Criteria:

* Must have had for at least 3 months painful diabetic neuropathy, or postherpetic neuralgia, or painful HIV-associated neuropathy, with moderate to severe pain on average.
* Must not have significant pain due to other causes (for example, arthritis).
* Must have intact skin at the treatment area.
* Must be prepared to remain on the same pain medications at the same doses as before the study for the entire duration of the study (12 weeks).
* Must not use topical pain medications on painful areas.
* Must be able to comply with study requirements such as completing daily pain diary and attending study visits and refrain from extensive travel during study participation.
* Must be at least 18 years old, not pregnant, and able to take care of self independently, with only occasional assistance if needed.
* No significant medical problems of the heart, kidneys, liver or lungs, or cancer.
* No history or current problem with substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - NeurogesX Investigational Site, Huntsville, Alabama
  - NeurogesX Investigational Site, Mobile, Alabama
  - NeurogesX Investigational Site, Phoenix, Arizona
  - NeurogesX Investigational Site, Fountain Valley, California
  - NeurogesX Investigational Site, Los Gatos, California
  - NeurogesX Investigational Site, Denver, Colorado
  - NeurogesX Investigational Site, Clearwater, Florida
  - NeurogesX Investigational Site, New Port Richey, Florida
  - NeurogesX Investigational Site, North Miami, Florida
  - NeurogesX Investigational Site, Plantation, Florida
  - NeurogesX Investigational Site, West Des Moines, Iowa
  - NeurogesX Investigational Site, Wellesley Hills, Massachusetts
  - NeurogesX Investigational Site, St Louis, Missouri
  - NeurogesX Investigational Site, Greensboro, New Jersey
  - NeurogesX Investigational Site, Duncansville, Pennsylvania
  - NeurogesX Investigational Site, San Antonio, Texas
  - NeurogesX Investigational Site, Salt Lake City, Utah

REFERENCES:
- [Derived] Webster LR, Peppin JF, Murphy FT, Lu B, Tobias JK, Vanhove GF. Efficacy, safety, and tolerability of NGX-4010, capsaicin 8% patch, in an open-label study of patients with peripheral neuropathic pain. Diabetes Res Clin Pract. 2011 Aug;93(2):187-197. doi: 10.1016/j.diabres.2011.04.010. Epub 2011 May 25. PMID 21612836